CLINICAL TRIAL: NCT02743585
Title: Impact of Rapid Pathogen Identification From Blood Cultures (RABbIT - Rapid Blood Culture Intervention Trial)
Brief Title: Impact of Rapid Pathogen Identification From Blood Cultures (RABbIT)
Acronym: RABbIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Shawn Vasoo, Consultant, Tan Tock Seng Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2015/00255
Record Dates: First submitted 2016-03-29; First posted 2016-04-19 (Estimated); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Bacteremia; Sepsis; Fungemia; Blood Stream Infection
MeSH Terms: conditions — Bacteremia; Sepsis; Fungemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Rapid diagnostic arm (Experimental): Standard Tan Tock Seng Hospital (TTSH) practices (bacterial culture and susceptibility testing) AND FilmArray Blood Culture ID (BCID) Panel test AND Rosco Diagnostica ESBL and carbapenemase screen will be performed.
  The Interventions to be administered are the rapid diagnostic tests: FilmArray Blood Culture ID (BCID) Panel test AND Rosco Diagnostica ESBL and carbapenemase screen.
  Subjects will be recruited 8am-3pm daily, weekdays only. Results of the BCID and Rosco test will be communicated to the managing physicians by phone in real-time.
  Interventions: Device: Filmarray Blood Culture ID (BCID) panel; Device: Rosco Diagnostica ESBL/carbapenemase screen kit
- Standard of care (control) (No Intervention): Standard Tan Tock Seng Hospital (TTSH) practices (bacterial culture and susceptibility testing) will be used. FilmArray BCID and Rosco Diagnostica ESBL and carbapenemase screen will NOT be performed. Subjects will be recruited 8am-3pm daily, weekdays only.

INTERVENTIONS:
Device: Filmarray Blood Culture ID (BCID) panel — The BCID panel is an FDA-approved nucleic acid amplification test (based on nested polymerase chain reaction) which detects Gram positive, Gram negative, the major Candida species and antimicrobial resistance markers (mecA for methicillin resistance, van A/B for vancomycin resistance, blaKPC for KPC carbapenemase) directly from positive blood cultures in < 1 - 1.5 hours
  Other Names: BCID
  Arms: Rapid diagnostic arm
Device: Rosco Diagnostica ESBL/carbapenemase screen kit — These kits are CE-marked (Approved in the European Union) rapid chromogenic tests for extended-spectrum beta-lactamase / carbapenemase detection from both blood cultures and cultured bacterial colonies.
  Arms: Rapid diagnostic arm

SUMMARY:
Septic shock carries high mortality, which may be exacerbated by inappropriate initial therapy. Inappropriate therapy may result from unanticipated antimicrobial resistance. Conversely, positive blood cultures may result from contamination, leading to unnecessary therapy and procedures and possibly prolonged hospitalization. Clinicians may also resort to broad spectrum antimicrobials and be hesitant to de-escalate while awaiting susceptibility results.

The investigators hypothesize that rapid identification of pathogens and antimicrobial resistance will ameliorate the above problems and improve time to optimal therapy, avoid unnecessary therapy and ultimately improve patient outcomes. While there are a number of in-vitro and uncontrolled clinical studies, there is a paucity of well-designed clinical trials objectively examining the real-world clinical and health-economic impact of such technology. To date only one randomised trial has been performed in the US (ClinicalTrials.gov NCT01898208), at a setting with low endemic rates of antimicrobial resistance. This is a companion study to NCT01898208. The investigators aim to study the clinical impact and cost-effectiveness of a strategy for rapid pathogen and resistance detection in a setting with a moderate to high levels of antimicrobial resistance.

DETAILED DESCRIPTION:
Hypothesis:

1. Rapid pathogen identification from blood cultures, including early identification of resistance (via specific genetic markers or phenotypic tests), will allow timelier initiation of appropriate antibiotic therapy and improved patient outcomes
2. Rapid organism identification from blood cultures will allow timelier initiation of effective and optimal antibiotic therapy; minimizing the use of unnecessary antibiotics, including combination therapy

Devices to be studied for this proposed study:

1. BCID panel (Biofire Diagnostics Inc., bioMerieux) : The BCID panel is an FDA-approved nucleic acid amplification test (based on nested polymerase chain reaction) which detects Gram positive, Gram negative, the major Candida species and antimicrobial resistance markers (mecA for methicillin resistance, van A/B for vancomycin resistance, blaKPC for Klebsiella pneumoniae carbapenemase (KPC)) directly from positive blood cultures in < 1 - 1.5 hours
2. Rosco Diagnostica extended-spectrum beta-lactamase (ESBL) and carbapenemase screen kit (Rosco Diagnostica): These kits are CE-marked (Approved in the European Union) rapid chromogenic tests for ESBL/ carbapenemase detection from both blood cultures and cultured bacterial colonies.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 21 years and above to 103 years
2. Blood culture flagged positive on automated instrument, with Gram positive, Gram negative bacteria or Yeast on Gram staining (including polymicrobial blood cultures)
3. Ability to provide informed consent or ability to obtain informed consent from legal guardian/representative (verbal and written)

Exclusion Criteria:

1. Patients whose blood cultures turn positive, but have no organism seen on Gram stain.
2. Patients who have been previously enrolled.
3. Patients who withdraw their consent (verbal or written).
4. Patients with any positive blood culture in the preceding 7 days.

Ages: 21 Years to 103 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 832 (Estimated)
Dates: Start 2017-03-20 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2020-07-02 (Estimated)

PRIMARY OUTCOMES:
Time from positive blood culture result to effective/optimal antibiotics | Approximately 14 days after positive blood culture
  An effective antibiotic is defined as an antibiotic regimen to which the bacterial/fungal isolate is susceptible (or predicted to be susceptible for Candida, per speciation).An optimal antibiotic is defined as an antibiotic regimen to which the bacterial/fungal isolate is susceptible/predicted to be susceptible, which is the most narrow spectrum and targeted, as recommended by institutional guidelines. This will be considered as the time from the positive Gram stain to first effective and the first optimal antibiotic.

SECONDARY OUTCOMES:
Clinical outcome (Infection related mortality) | 1 year
  Infection-related at 30-day, 90-days and 1-year
Clinical outcome (All-cause related mortality) | 1 year
  All cause mortality at 30-day, 90-days and 1-year mortality
Clinical outcome (Quality of life) | 1 year
  Quality of life at enrolment, 90-days and at 1 year, as measured by the tools EQ-5D-5L QoL/SF-12
Time from positive blood culture result to bacterial identification | Approximately 3 days
Duration of hospitalization (days) | Participants were followed for the duration of hospital stay, approximately 28 days
Duration of bacteremia/fungemia (days) | Patient-dependent variable, estimated up to 7 days
Time to isolation precautions | Estimated up to 5 days
  Time taken for implementation of appropriate infection control measures (isolation precautions) as appropriate for pathogen detected
Antibiotic-associated adverse events | Approximately 14 days after positive blood culture
  This included all adverse events that occurred within 2 weeks following enrollment and were documented in the medical record.
Antimicrobial utilization (hours/days of therapy) | Approximately 4 days after enrollment
  Difference between the date and time of the antibiotic start order (or Gram stain-positive blood culture, if antibiotics were started prior to the positive culture result) and the date and time of the antibiotic stop order. Shorter duration of broad spectrum antibiotics and longer duration of narrow-spectrum antibiotics were considered favorable outcomes.
Mean Total Hospitalization Costs Per Subject | Approximately 7 days after positive blood culture for up to an estimated 24 weeks
  These will be calculated based on actual billable patient costs (without government subventions/subsidies) following 7 days after the positive blood culture episode and for the duration of hospitalization, up to an estimated 24 weeks.
Mean Laboratory Costs Per Subject | Approximately 7 days after positive blood culture for up to an estimated 24 week
  These will be calculated based on actual billable laboratory costs (without government subventions/subsidies) following 7 days after the positive blood culture episode and for the duration of hospitalization, up to an estimated 24 weeks.
Mean Antimicrobials Costs Per Subject | Approximately 7 days after positive blood culture and for duration of entire hospitalization
  These will be calculated based on actual billable antimicrobial costs (without government subventions/subsidies) following 7 days after the positive blood culture episode and for the duration of hospitalization, up to an estimated 24 weeks.
Cost-effectiveness analysis | Up to 1 year after enrolment and using a 'modeled horizon' based on sepsis-adjusted life expectancies
  Incremental cost-effectiveness ratios will be determined by dividing the difference between the average costs of treating a patient in the after phase (C1) and the average cost in the before phase (C0) by the difference between average health outcomes (QALYs) gained in the after phase (O1) and those gained in the before phase (O0). The incremental cost-effectiveness ratio is calculated by the following equation: (C1 - C0)/(O1 - O0). Incremental cost-effectiveness ratios using quality adjusted/sepsis adjusted life years gained as the health outcome of interest will then be determined, based on the method of Jones et al Crit Care Med. 2011 June ; 39(6): 1306-1312.
Time on effective/optimal antibiotics within first 96 hours of positive blood culture | First 96 hours after blood culture turns positive
  An effective antibiotic is defined as an antibiotic regimen to which the bacterial/fungal isolate is susceptible (or predicted to be susceptible for Candida, per speciation).An optimal antibiotic is defined as an antibiotic regimen to which the bacterial/fungal isolate is susceptible/predicted to be susceptible, which is the most narrow spectrum and targeted, as recommended by institutional guidelines. This will be considered in the 96-hour time frame from the positive Gram stain.

OTHER OUTCOMES:
Time to First Appropriate De-escalation or First Appropriate Escalation of Antibiotics | Positive Gram stain, 96 hours after enrollment
  De-escalation included discontinuation of 1 or more antibiotics and/or switching from a broad- to a narrow spectrum antibiotic. Escalation included initiation of 1 or more antibiotics and/or switching from a narrow- to a broad-spectrum antibiotic
Percent of Contaminated Blood Cultures Not Treated or Treated for Less Than 24 Hours | Within 24 hours after positive blood culture
  Contaminated blood cultures were defined as growth of organisms such as coagulase-negative staphylococci from a single blood culture set when greater than or equal to 2 blood culture sets were collected, except among subjects suspected to have true bacteremia associated with central venous catheters or devices.
Length of Entire Hospitalization (Days) | Participants are followed for the duration of hospital stay, approximately 15 days
Percentage of Subjects With Infectious Disease Consultation Within 72 Hours of Enrollment | Approximately within 72 hours of positive blood culture
Length of Intensive Care Unit Stay (days) | Within 14 days of positive blood culture until ICU discharge, up to an estimated 24 weeks.
Percentage of Patients Who Acquired Clostridium Difficile Within 30 Days After Enrollment | Approximately 30 days after positive blood culture
Percentage of Patients Who Acquired Multidrug-resistant organisms Within 30 Days After Enrollment | Approximately 30 days after positive blood culture
  Multidrug-resistant organisms included vancomycin-resistant enterococci, methicillin-resistant Staphylococcus aureus, extended-spectrum cephalosporin-resistant Enterobacteriaceae, and Pseudomonas aeruginosa and Acinetobacter species resistant to greater than or equal to 3 antibiotic classes.

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Vasoo, MD, Principal Investigator — Tan Tock Seng Hospital; Partha P De, MD, Principal Investigator — Tan Tock Seng Hospital; Christine B Teng, MSc, Principal Investigator — National University of Singapore/Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ong SWX, Hon PY, Wee SSH, Chia JWZ, Mendis S, Izharuddin E, Lin RJ, Chia PY, Sim RCS, Chen MI, Chow A, Yoong J, Lye DC, Teng CB, Tambyah PA, Banerjee R, Patel R, De PP, Vasoo S. Accuracy of a Rapid Multiplex Polymerase Chain Reaction Plus a Chromogenic Phenotypic Test Algorithm for Detection of Extended-Spectrum beta-Lactamase and Carbapenemase-Producing Gram-Negative Bacilli in Positive Blood Culture Bottles. Clin Infect Dis. 2022 May 30;74(10):1850-1854. doi: 10.1093/cid/ciab848. PMID 34554228